CLINICAL TRIAL: NCT06864403
Title: Mirikizumab in the Treatment of Chronic Inflammatory Conditions of the Pouch
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-2214
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-09

CONDITIONS: Pouchitis; Pouches, Ileoanal; Pouch, Ileal
Keywords: mirikizumab; Omvoh; chronic pouchitis; IPAA; Crohn's-like disease of the pouch; Ileal Pouch Anal Anastomosis
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Intervention Model Description: Interventional Study, open-label real-world observational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Other): Open Label Mirikizumab
  Interventions: Drug: Mirikizumab - Intravenous (IV); Drug: Mirikizumab - Subcutaneous (SC)

INTERVENTIONS:
Drug: Mirikizumab - Intravenous (IV) — 300 mg mirikizumab at Weeks 0, 4, and 8
  Other Names: Omvoh
Drug: Mirikizumab - Subcutaneous (SC) — Pre-filled syringes administered at Weeks 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52.
  Other Names: Omvoh

SUMMARY:
The goal of this clinical trial is to learn if mirikizumab works to treat pouch disorders in adults. The main questions it aims to answer are:

Does mirikizumab reduce symptoms of pouch disorders

Participants will:

Take mirikizumab every 4 weeks for one year Visit the clinic once every month for two months and at the end of the study Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained before any study-related procedures
* Age >/= 18 and </= 80 years
* Diagnosis of Chronic Pouchitis or Crohn's-like disease of the pouch based on the following criteria:

  * Chronic Antibiotic-Dependent Pouchitis: Recurrent symptoms of pouchitis (frequency, urgency, bleeding, abdominal pain or cramping, or pelvic discomfort) that respond to antibiotic therapy but relapse shortly after stopping antibiotics, thus necessitating continuous antibiotic therapy to achieve symptom control.
  * Chronic Antibiotic Refractory Pouchitis: Lack of response to standard antibiotic therapy, requirement of a longer duration of antibiotic therapy than expected with minimal improvement in symptoms, in association with typical symptoms of pouchitis (frequency, urgency, bleeding, abdominal pain or cramping, or pelvic discomfort).
  * Crohn's-like disease of the pouch: Presence of a perianal or other fistula that developed at least 12 months after the final stage of Ileal Pouch Anal Anastomosis (IPAA) surgery, stricture of the pouch body or pre-pouch ileum, or the presence of pre-pouch ileitis. Pouch body inflammation (pouchitis) may often coexist in the setting of Crohn's-like disease of the pouch.
* Participants with a proven history of ulcerative colitis and history of 1,2, modified -2 or 3 stage IPAA and ileostomy takedown
* Ability to access internet for electronic database entry
* Only those individuals for whom a provider is considering initiating mirikizumab for the treatment of chronic pouchitis or Crohn's-like disease of the pouch will be eligible for participation.

Exclusion Criteria:

* Prior exposure to mirikizumab
* Known hypersensitivity to mirikizumab or its metabolites
* Current infection with Clostridioides difficile
* Known HIV or active Hepatitis B/C
* Clinically significant liver disease (Primary Sclerosing Cholangitis with LFT's <1.5 upper limit of normal can be included)
* Severe hepatic impairment, defined as Child-Pugh Class C
* Known decreased kidney function with a glomerular filtration rate <45 ml/min/1.732
* History of malignancy, except for basal cell carcinoma, non-metastatic squamous cell carcinoma of the skin, or prior malignancy with curative therapy completed at least 5 years prior to screening and no recurrence.
* Clinically significant laboratory results at screening or baseline, as judged by the Investigator from local testing.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using a highly effective contraceptive method.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening.
* Any disorder, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Remission as measured by Modified Pouchitis Disease Activity Index (mPDAI) | Weeks 0, 24, and 52
  The Pouchitis Disease Activity Index (PDAI) was developed for diagnosing active pouchitis and quantifying the severity of pouchitis. The PDAI includes the clinical criteria of 1) stool frequency 2) rectal bleeding 3) Fecal Urgency/Abdominal Cramps and 4) presence or absence of fever, endoscopic criteria, and histologic criteria through biopsies. The PDAI was modified to omit the biopsy and histology costs. The mPDAI includes the clinical portion and the endoscopic subscore of the PDAI. Score range is 0-12. The higher the score, the worse the disease activity. mPDAI remission is defined as an mPDAI score of 4 or lower and a reduction from baseline of 2 or more points in the mPDAI total score.

SECONDARY OUTCOMES:
Median change in the Endoscopic Pouch Score (EPS) | Weeks 0, 24, and 52
  The endoscopic pouch score (EPS) is a standardized assessment of inflammation in the pouch of patients with an ileal pouch anal anastomosis (IPAA), including those with inflammation outside the pouch body. The EPS is a novel method of endoscopic scoring that has been developed to offer more granular longitudinal assessments of response to advanced therapies in patients with inflammatory conditions of the pouch. Score range is 0-45. The higher the score, the worse the disease activity.
Median change in the endoscopic subscore of the mPDAI | Weeks 0, 24, and 52
  The endoscopic subscore of the PDAI is a component of the PDAI that assesses endoscopic findings of pouchitis. Score range is 0-6. The higher the score, the worse the disease activity.
Change in Cleveland Clinic Global Quality of Life (QoL) scale | Weeks 0, 4, 8, 12, 24, 38, and 52
  The Cleveland Clinic Global Quality of Life scale asks the patient to rate their current QoL, current quality of health, and current energy level using a 1-10 rating (where 10 is best). The score on each of these 3 components is added and the final Cleveland Clinic Global Quality of Life utility score can be obtained by dividing this result by 30. A higher score means improved quality of life.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) incontinence measures | Weeks 0, 4, 8, 12, 24, 38, and 52
  The PROMIS measure for incontinence includes 4 items that assess the frequency of bowel incontinence, soiling, stool leakage, and stool leakage while passing gas over the past 7 days. Score range is 0-20, where a higher score means increased incontinence.
Change in Urgency Numeric Rating Scale (NRS) | Weeks 0, 4, 8, 12, 24, 38, and 52
  Urgency will be measured by the 11-point Likert scale urgency question as validated in the mirikizumab clinical trials. Score range is 0-10. The higher the score, the worse the urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Barnes, MD, MPH, Principal Investigator — University of North Carolina
Locations (5):
- United States (5):
  - UCLA Vatche & Tamar Manoukian Division of Digestive Diseases, Los Angeles, California
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 12 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning 9 and continuing for 12 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Weaver KN, Gregory M, Syal G, Hoversten P, Hicks SB, Patel D, Christophi G, Beniwal-Patel P, Isaacs KL, Raffals L, Deepak P, Herfarth HH, Barnes EL. Ustekinumab Is Effective for the Treatment of Crohn's Disease of the Pouch in a Multicenter Cohort. Inflamm Bowel Dis. 2019 Mar 14;25(4):767-774. doi: 10.1093/ibd/izy302. PMID 30295784
- [Background] Gregory M, Weaver KN, Hoversten P, Hicks SB, Patel D, Ciorba MA, Gutierrez AM, Beniwal-Patel P, Palam S, Syal G, Herfarth HH, Christophi G, Raffals L, Barnes EL, Deepak P. Efficacy of Vedolizumab for Refractory Pouchitis of the Ileo-anal Pouch: Results From a Multicenter US Cohort. Inflamm Bowel Dis. 2019 Aug 20;25(9):1569-1576. doi: 10.1093/ibd/izz030. PMID 30810748
- [Background] Ollech JE, Rubin DT, Glick L, Weisshof R, El Jurdi K, Israel A, Krugliak Cleveland N, Hyman N, Sakuraba A, Pekow J, Cohen RD, Dalal SR. Ustekinumab Is Effective for the Treatment of Chronic Antibiotic-Refractory Pouchitis. Dig Dis Sci. 2019 Dec;64(12):3596-3601. doi: 10.1007/s10620-019-05697-1. Epub 2019 Jun 11. PMID 31187322
- [Background] Akiyama S, Cohen NA, Kayal M, Dubinsky MC, Colombel JF, Rubin DT. Treatment of Chronic Inflammatory Pouch Conditions With Tofacitinib: A Case Series From 2 Tertiary IBD Centers in the United States. Inflamm Bowel Dis. 2023 Sep 1;29(9):1504-1507. doi: 10.1093/ibd/izad011. No abstract available. PMID 36745039
- [Background] Kayal M, Lambin T, Plietz M, Rizvi A, Radcliffe M, Khaitov S, Sylla P, Greenstein AJ, Colombel JF, Dubinsky MC, Ungaro RC. Recycling of Precolectomy Anti-Tumor Necrosis Factor Agents in Chronic Pouch Inflammation Is Associated With Treatment Failure. Clin Gastroenterol Hepatol. 2021 Jul;19(7):1491-1493.e3. doi: 10.1016/j.cgh.2020.07.008. Epub 2020 Jul 12. PMID 32668342
- [Background] Shen B, Achkar JP, Connor JT, Ormsby AH, Remzi FH, Bevins CL, Brzezinski A, Bambrick ML, Fazio VW, Lashner BA. Modified pouchitis disease activity index: a simplified approach to the diagnosis of pouchitis. Dis Colon Rectum. 2003 Jun;46(6):748-53. doi: 10.1007/s10350-004-6652-8. PMID 12794576
- [Background] Barnes EL, Long MD, Raffals L, Isaacs K, Stidham RW, Herfarth HH; Contributors. Development of the Endoscopic Pouch Score for Assessment of Inflammatory Conditions of the Pouch. Clin Gastroenterol Hepatol. 2023 Jun;21(6):1663-1666.e3. doi: 10.1016/j.cgh.2022.04.026. Epub 2022 May 12. PMID 35568303
- [Background] Dubinsky MC, Irving PM, Panaccione R, Naegeli AN, Potts-Bleakman A, Arora V, Shan M, Travis S. Incorporating patient experience into drug development for ulcerative colitis: development of the Urgency Numeric Rating Scale, a patient-reported outcome measure to assess bowel urgency in adults. J Patient Rep Outcomes. 2022 Apr 1;6(1):31. doi: 10.1186/s41687-022-00439-w. PMID 35362902
- [Background] Yamamoto T, Shimoyama T, Bamba T, Matsumoto K. Consecutive Monitoring of Fecal Calprotectin and Lactoferrin for the Early Diagnosis and Prediction of Pouchitis after Restorative Proctocolectomy for Ulcerative Colitis. Am J Gastroenterol. 2015 Jun;110(6):881-7. doi: 10.1038/ajg.2015.129. Epub 2015 Apr 28. PMID 25916224
- [Background] Lin JF, Chen JM, Zuo JH, Yu A, Xiao ZJ, Deng FH, Nie B, Jiang B. Meta-analysis: fecal calprotectin for assessment of inflammatory bowel disease activity. Inflamm Bowel Dis. 2014 Aug;20(8):1407-15. doi: 10.1097/MIB.0000000000000057. PMID 24983982
- [Background] Ollech JE, Bannon L, Maharshak N, Bar N, Goren I, Tulchinsky H, Yanai H, Dotan I. Fecal Calprotectin Is Increased in Pouchitis and Progressively Increases With More Severe Endoscopic and Histologic Disease. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1839-1846.e2. doi: 10.1016/j.cgh.2021.11.012. Epub 2021 Nov 16. PMID 34798336
- [Background] Singh S, Ananthakrishnan AN, Nguyen NH, Cohen BL, Velayos FS, Weiss JM, Sultan S, Siddique SM, Adler J, Chachu KA; AGA Clinical Guidelines Committee. Electronic address: clinicalpractice@gastro.org. AGA Clinical Practice Guideline on the Role of Biomarkers for the Management of Ulcerative Colitis. Gastroenterology. 2023 Mar;164(3):344-372. doi: 10.1053/j.gastro.2022.12.007. PMID 36822736
- [Background] Fazio VW, O'Riordain MG, Lavery IC, Church JM, Lau P, Strong SA, Hull T. Long-term functional outcome and quality of life after stapled restorative proctocolectomy. Ann Surg. 1999 Oct;230(4):575-84; discussion 584-6. doi: 10.1097/00000658-199910000-00013. PMID 10522727
- [Background] D'Haens G, Dubinsky M, Kobayashi T, Irving PM, Howaldt S, Pokrotnieks J, Krueger K, Laskowski J, Li X, Lissoos T, Milata J, Morris N, Arora V, Milch C, Sandborn W, Sands BE; LUCENT Study Group. Mirikizumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2023 Jun 29;388(26):2444-2455. doi: 10.1056/NEJMoa2207940. PMID 37379135
- [Background] Sands BE, D'Haens G, Clemow DB, Irving PM, Johns JT, Hunter Gibble T, Abreu MT, Lee S, Hisamatsu T, Kobayashi T, Dubinsky MC, Vermeire S, Siegel CA, Peyrin-Biroulet L, Moses RE, Milata J, Arora V, Panaccione R, Dignass A. Two-Year Efficacy and Safety of Mirikizumab Following 104 Weeks of Continuous Treatment for Ulcerative Colitis: Results From the LUCENT-3 Open-Label Extension Study. Inflamm Bowel Dis. 2024 Dec 5;30(12):2245-2258. doi: 10.1093/ibd/izae024. PMID 38459910
- [Background] Devaraj B, Kaiser AM. Surgical management of ulcerative colitis in the era of biologicals. Inflamm Bowel Dis. 2015 Jan;21(1):208-20. doi: 10.1097/MIB.0000000000000178. PMID 25222665
- [Background] Barnes EL, Herfarth HH, Kappelman MD, Zhang X, Lightner A, Long MD, Sandler RS. Incidence, Risk Factors, and Outcomes of Pouchitis and Pouch-Related Complications in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2021 Aug;19(8):1583-1591.e4. doi: 10.1016/j.cgh.2020.06.035. Epub 2020 Jun 22. PMID 32585362
- [Background] Barnes EL, Jiang Y, Kappelman MD, Long MD, Sandler RS, Kinlaw AC, Herfarth HH. Decreasing Colectomy Rate for Ulcerative Colitis in the United States Between 2007 and 2016: A Time Trend Analysis. Inflamm Bowel Dis. 2020 Jul 17;26(8):1225-1231. doi: 10.1093/ibd/izz247. PMID 31634390
- [Background] Bertucci Zoccali M, Hyman NH, Skowron KB, Rubin M, Cannon LM, Hurst RD, Umanskiy K, Rubin DT, Shogan BD. Exposure to Anti-tumor Necrosis Factor Medications Increases the Incidence of Pouchitis After Restorative Proctocolectomy in Patients With Ulcerative Colitis. Dis Colon Rectum. 2019 Nov;62(11):1344-1351. doi: 10.1097/DCR.0000000000001467. PMID 31596761
- [Background] Barnes EL, Allin KH, Iversen AT, Herfarth HH, Jess T. Increasing Incidence of Pouchitis Between 1996 and 2018: A Population-Based Danish Cohort Study. Clin Gastroenterol Hepatol. 2023 Jan;21(1):192-199.e7. doi: 10.1016/j.cgh.2022.04.015. Epub 2022 May 5. PMID 35525393
- [Background] Barnes EL, Herfarth HH, Sandler RS, Chen W, Jaeger E, Nguyen VM, Robb AR, Kappelman MD, Martin CF, Long MD. Pouch-Related Symptoms and Quality of Life in Patients with Ileal Pouch-Anal Anastomosis. Inflamm Bowel Dis. 2017 Jul;23(7):1218-1224. doi: 10.1097/MIB.0000000000001119. PMID 28426474
- [Background] Barnes EL, Kappelman MD, Zhang X, Long MD, Sandler RS, Herfarth HH. Patients With Pouchitis Demonstrate a Significant Cost Burden in the First Two Years After Ileal Pouch-Anal Anastomosis. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2908-2910.e2. doi: 10.1016/j.cgh.2021.09.037. Epub 2021 Oct 2. PMID 34610443
- [Background] Fazio VW, Kiran RP, Remzi FH, Coffey JC, Heneghan HM, Kirat HT, Manilich E, Shen B, Martin ST. Ileal pouch anal anastomosis: analysis of outcome and quality of life in 3707 patients. Ann Surg. 2013 Apr;257(4):679-85. doi: 10.1097/SLA.0b013e31827d99a2. PMID 23299522
- [Background] Barnes EL, Kochar B, Jessup HR, Herfarth HH. The Incidence and Definition of Crohn's Disease of the Pouch: A Systematic Review and Meta-analysis. Inflamm Bowel Dis. 2019 Aug 20;25(9):1474-1480. doi: 10.1093/ibd/izz005. PMID 30698715
- [Background] Barnes EL, Agrawal M, Syal G, Ananthakrishnan AN, Cohen BL, Haydek JP, Al Kazzi ES, Eisenstein S, Hashash JG, Sultan SS, Raffals LE, Singh S; AGA Clinical Guidelines Committee. Electronic address: clinicalpractice@gastro.org. AGA Clinical Practice Guideline on the Management of Pouchitis and Inflammatory Pouch Disorders. Gastroenterology. 2024 Jan;166(1):59-85. doi: 10.1053/j.gastro.2023.10.015. PMID 38128971
- [Background] Kayal M, Deepak P, Beniwal-Patel P, Raffals L, Dubinsky M, Chang S, Higgins PDR, Jiang Y, Cross RK, Long MD, Herfarth HH, Barnes EL. Changes in Therapy Are Not Associated With Increased Remission in Patients With Crohn's Disease of the Pouch. Am J Gastroenterol. 2024 Mar 1;119(3):584-587. doi: 10.14309/ajg.0000000000002599. Epub 2023 Nov 17. PMID 37975591
- [Background] Barnes EL, Deepak P, Beniwal-Patel P, Raffals L, Kayal M, Dubinsky M, Chang S, Higgins PDR, Barr JI, Galanko J, Jiang Y, Cross RK, Long MD, Herfarth HH. Treatment Patterns and Standardized Outcome Assessments Among Patients With Inflammatory Conditions of the Pouch in a Prospective Multicenter Registry. Crohns Colitis 360. 2022 Aug 2;4(3):otac030. doi: 10.1093/crocol/otac030. eCollection 2022 Jul. PMID 36082341
- [Background] Batista D, Raffals L. Role of intestinal bacteria in the pathogenesis of pouchitis. Inflamm Bowel Dis. 2014 Aug;20(8):1481-6. doi: 10.1097/MIB.0000000000000055. PMID 25046009
- [Background] Lovegrove RE, Tilney HS, Heriot AG, von Roon AC, Athanasiou T, Church J, Fazio VW, Tekkis PP. A comparison of adverse events and functional outcomes after restorative proctocolectomy for familial adenomatous polyposis and ulcerative colitis. Dis Colon Rectum. 2006 Sep;49(9):1293-306. doi: 10.1007/s10350-006-0608-0. PMID 16830218
- [Background] Shen B, Lashner B. Can we immunogenotypically and immunophenotypically profile patients who are at risk for pouchitis? Am J Gastroenterol. 2004 Mar;99(3):442-4. doi: 10.1111/j.1572-0241.2004.04096.x. No abstract available. PMID 15056082
- [Background] Meier CB, Hegazi RA, Aisenberg J, Legnani PE, Nilubol N, Cobrin GM, Duerr RH, Gorfine SR, Bauer JJ, Sachar DB, Plevy SE. Innate immune receptor genetic polymorphisms in pouchitis: is CARD15 a susceptibility factor? Inflamm Bowel Dis. 2005 Nov;11(11):965-71. doi: 10.1097/01.mib.0000186407.25694.cf. PMID 16239841
- [Background] Tyler AD, Milgrom R, Stempak JM, Xu W, Brumell JH, Muise AM, Sehgal R, Cohen Z, Koltun W, Shen B, Silverberg MS. The NOD2insC polymorphism is associated with worse outcome following ileal pouch-anal anastomosis for ulcerative colitis. Gut. 2013 Oct;62(10):1433-9. doi: 10.1136/gutjnl-2011-301957. Epub 2012 Aug 9. PMID 22879519
- [Background] Carter MJ, Di Giovine FS, Cox A, Goodfellow P, Jones S, Shorthouse AJ, Duff GW, Lobo AJ. The interleukin 1 receptor antagonist gene allele 2 as a predictor of pouchitis following colectomy and IPAA in ulcerative colitis. Gastroenterology. 2001 Oct;121(4):805-11. doi: 10.1053/gast.2001.28017. PMID 11606494
- [Background] Lammers KM, Ouburg S, Morre SA, Crusius JB, Gionchett P, Rizzello F, Morselli C, Caramelli E, Conte R, Poggioli G, Campieri M, Pena AS. Combined carriership of TLR9-1237C and CD14-260T alleles enhances the risk of developing chronic relapsing pouchitis. World J Gastroenterol. 2005 Dec 14;11(46):7323-9. doi: 10.3748/wjg.v11.i46.7323. PMID 16437636
- [Background] Lim M, Adams JD, Wilcox M, Finan P, Sagar P, Burke D. An assessment of bacterial dysbiosis in pouchitis using terminal restriction fragment length polymorphisms of 16S ribosomal DNA from pouch effluent microbiota. Dis Colon Rectum. 2009 Aug;52(8):1492-500. doi: 10.1007/DCR.0b013e3181a7b77a. PMID 19617766
- [Background] Coffey JC, Rowan F, Burke J, Dochery NG, Kirwan WO, O'Connell PR. Pathogenesis of and unifying hypothesis for idiopathic pouchitis. Am J Gastroenterol. 2009 Apr;104(4):1013-23. doi: 10.1038/ajg.2008.127. Epub 2009 Mar 3. PMID 19259080
- [Background] Sokol H, Lay C, Seksik P, Tannock GW. Analysis of bacterial bowel communities of IBD patients: what has it revealed? Inflamm Bowel Dis. 2008 Jun;14(6):858-67. doi: 10.1002/ibd.20392. PMID 18275077
- [Background] Komanduri S, Gillevet PM, Sikaroodi M, Mutlu E, Keshavarzian A. Dysbiosis in pouchitis: evidence of unique microfloral patterns in pouch inflammation. Clin Gastroenterol Hepatol. 2007 Mar;5(3):352-60. doi: 10.1016/j.cgh.2007.01.001. PMID 17368235
- [Background] Dubinsky V, Reshef L, Bar N, Keizer D, Golan N, Rabinowitz K, Godny L, Yadgar K, Zonensain K, Tulchinsky H, Gophna U, Dotan I. Predominantly Antibiotic-resistant Intestinal Microbiome Persists in Patients With Pouchitis Who Respond to Antibiotic Therapy. Gastroenterology. 2020 Feb;158(3):610-624.e13. doi: 10.1053/j.gastro.2019.10.001. Epub 2019 Oct 9. PMID 31605691
- [Background] Duffy M, O'Mahony L, Coffey JC, Collins JK, Shanahan F, Redmond HP, Kirwan WO. Sulfate-reducing bacteria colonize pouches formed for ulcerative colitis but not for familial adenomatous polyposis. Dis Colon Rectum. 2002 Mar;45(3):384-8. doi: 10.1007/s10350-004-6187-z. PMID 12068199
- [Background] Smith FM, Coffey JC, Kell MR, O'Sullivan M, Redmond HP, Kirwan WO. A characterization of anaerobic colonization and associated mucosal adaptations in the undiseased ileal pouch. Colorectal Dis. 2005 Nov;7(6):563-70. doi: 10.1111/j.1463-1318.2005.00833.x. PMID 16232236
- [Background] Machiels K, Sabino J, Vandermosten L, Joossens M, Arijs I, de Bruyn M, Eeckhaut V, Van Assche G, Ferrante M, Verhaegen J, Van Steen K, Van Immerseel F, Huys G, Verbeke K, Wolthuis A, de Buck Van Overstraeten A, D'Hoore A, Rutgeerts P, Vermeire S. Specific members of the predominant gut microbiota predict pouchitis following colectomy and IPAA in UC. Gut. 2017 Jan;66(1):79-88. doi: 10.1136/gutjnl-2015-309398. Epub 2015 Sep 30. PMID 26423113
- [Background] Atarashi K, Suda W, Luo C, Kawaguchi T, Motoo I, Narushima S, Kiguchi Y, Yasuma K, Watanabe E, Tanoue T, Thaiss CA, Sato M, Toyooka K, Said HS, Yamagami H, Rice SA, Gevers D, Johnson RC, Segre JA, Chen K, Kolls JK, Elinav E, Morita H, Xavier RJ, Hattori M, Honda K. Ectopic colonization of oral bacteria in the intestine drives TH1 cell induction and inflammation. Science. 2017 Oct 20;358(6361):359-365. doi: 10.1126/science.aan4526. PMID 29051379
- [Background] Travis S, Silverberg MS, Danese S, Gionchetti P, Lowenberg M, Jairath V, Feagan BG, Bressler B, Ferrante M, Hart A, Lindner D, Escher A, Jones S, Shen B; EARNEST Study Group. Vedolizumab for the Treatment of Chronic Pouchitis. N Engl J Med. 2023 Mar 30;388(13):1191-1200. doi: 10.1056/NEJMoa2208450. PMID 36988594
- [Background] Chandan S, Mohan BP, Kumar A, Khan SR, Chandan OC, Kassab LL, Ponnada S, Kochhar GS. Safety and Efficacy of Biological Therapy in Chronic Antibiotic Refractory Pouchitis: A Systematic Review With Meta-analysis. J Clin Gastroenterol. 2021 Jul 1;55(6):481-491. doi: 10.1097/MCG.0000000000001550. PMID 34049383
- [Background] Herfarth HH, Long MD, Isaacs KL. Use of Biologics in Pouchitis: A Systematic Review. J Clin Gastroenterol. 2015 Sep;49(8):647-54. doi: 10.1097/MCG.0000000000000367. PMID 26084005
- [Background] Sandborn WJ, Ferrante M, Bhandari BR, Berliba E, Feagan BG, Hibi T, Tuttle JL, Klekotka P, Friedrich S, Durante M, Morgan-Cox M, Laskowski J, Schmitz J, D'Haens GR. Efficacy and Safety of Mirikizumab in a Randomized Phase 2 Study of Patients With Ulcerative Colitis. Gastroenterology. 2020 Feb;158(3):537-549.e10. doi: 10.1053/j.gastro.2019.08.043. Epub 2019 Sep 4. PMID 31493397
- [Background] Kochar B, Martin CF, Kappelman MD, Spiegel BM, Chen W, Sandler RS, Long MD. Evaluation of Gastrointestinal Patient Reported Outcomes Measurement Information System (GI-PROMIS) Symptom Scales in Subjects With Inflammatory Bowel Diseases. Am J Gastroenterol. 2018 Jan;113(1):72-79. doi: 10.1038/ajg.2017.240. Epub 2017 Aug 29. PMID 28853727
- [Background] Sandborn WJ, Tremaine WJ, Batts KP, Pemberton JH, Phillips SF. Pouchitis after ileal pouch-anal anastomosis: a Pouchitis Disease Activity Index. Mayo Clin Proc. 1994 May;69(5):409-15. doi: 10.1016/s0025-6196(12)61634-6. PMID 8170189
- [Background] Isaacs KL, Sandler RS, Abreu M, Picco MF, Hanauer SB, Bickston SJ, Present D, Farraye FA, Wolf D, Sandborn WJ; Crohn's and Colitis Foundation of America Clinical Alliance. Rifaximin for the treatment of active pouchitis: a randomized, double-blind, placebo-controlled pilot study. Inflamm Bowel Dis. 2007 Oct;13(10):1250-5. doi: 10.1002/ibd.20187. PMID 17567869
- [Background] Gionchetti P, Morselli C, Rizzello F, et al. Infliximab in the treatment of refractory pouchitis. Gastroenterology 2005;128:A578-A578
- [Background] Gionchetti P, Rizzello F, Helwig U, Venturi A, Lammers KM, Brigidi P, Vitali B, Poggioli G, Miglioli M, Campieri M. Prophylaxis of pouchitis onset with probiotic therapy: a double-blind, placebo-controlled trial. Gastroenterology. 2003 May;124(5):1202-9. doi: 10.1016/s0016-5085(03)00171-9. PMID 12730861
- [Background] Gionchetti P, Rizzello F, Morselli C, Poggioli G, Tambasco R, Calabrese C, Brigidi P, Vitali B, Straforini G, Campieri M. High-dose probiotics for the treatment of active pouchitis. Dis Colon Rectum. 2007 Dec;50(12):2075-82; discussion 2082-4. doi: 10.1007/s10350-007-9068-4. Epub 2007 Oct 13. PMID 17934776
- [Background] Gionchetti P, Rizzello F, Venturi A, Brigidi P, Matteuzzi D, Bazzocchi G, Poggioli G, Miglioli M, Campieri M. Oral bacteriotherapy as maintenance treatment in patients with chronic pouchitis: a double-blind, placebo-controlled trial. Gastroenterology. 2000 Aug;119(2):305-9. doi: 10.1053/gast.2000.9370. PMID 10930365
- [Background] Gionchetti P, Rizzello F, Venturi A, Ugolini F, Rossi M, Brigidi P, Johansson R, Ferrieri A, Poggioli G, Campieri M. Antibiotic combination therapy in patients with chronic, treatment-resistant pouchitis. Aliment Pharmacol Ther. 1999 Jun;13(6):713-8. doi: 10.1046/j.1365-2036.1999.00553.x. PMID 10383499
- [Background] Kuhbacher T, Ott SJ, Helwig U, Mimura T, Rizzello F, Kleessen B, Gionchetti P, Blaut M, Campieri M, Folsch UR, Kamm MA, Schreiber S. Bacterial and fungal microbiota in relation to probiotic therapy (VSL#3) in pouchitis. Gut. 2006 Jun;55(6):833-41. doi: 10.1136/gut.2005.078303. Epub 2006 Jan 9. PMID 16401690
- [Background] Mimura T, Rizzello F, Helwig U, Poggioli G, Schreiber S, Talbot IC, Nicholls RJ, Gionchetti P, Campieri M, Kamm MA. Once daily high dose probiotic therapy (VSL#3) for maintaining remission in recurrent or refractory pouchitis. Gut. 2004 Jan;53(1):108-14. doi: 10.1136/gut.53.1.108. PMID 14684584
- [Background] Shen B, Remzi FH, Lopez AR, Queener E. Rifaximin for maintenance therapy in antibiotic-dependent pouchitis. BMC Gastroenterol. 2008 Jun 23;8:26. doi: 10.1186/1471-230X-8-26. PMID 18573211
- [Background] Barnes EL, Boynton MH, DeWalt DA, Herfarth HH, Kappelman MD. Patient Reported Outcome Assessments Used in the Evaluation of Patients after Ileal Pouch-Anal Anastomosis: A Systematic Review. Gastro Hep Adv. 2023;2(8):1044-1049. doi: 10.1016/j.gastha.2023.07.010. Epub 2023 Jul 29. PMID 38125203
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Background] Dubinsky MC, Panaccione R, Lewis JD, Sands BE, Hibi T, Lee SD, Naegeli AN, Shan M, Green LA, Morris N, Arora V, Bleakman AP, Belin R, Travis S. Impact of Bowel Urgency on Quality of Life and Clinical Outcomes in Patients With Ulcerative Colitis. Crohns Colitis 360. 2022 Jun 3;4(3):otac016. doi: 10.1093/crocol/otac016. eCollection 2022 Jul. PMID 36777426
- [Background] Barnes EL. A Practical Guide to the Use of Mirikizumab. Am J Gastroenterol. 2024 Mar 1;119(3):400-403. doi: 10.14309/ajg.0000000000002531. Epub 2023 Oct 2. No abstract available. PMID 37782274
- [Background] European Medicines Agency: Vedolizumab.